CLINICAL TRIAL: NCT06143735
Title: A Randomized, Multicenter, Exploratory Clinical Study for The Primary And Secondary Prevention of Febrile Neutropenia (FN) With Efbemalenograstim Alfa in Patients With Non-small Cell Lung Cancer (NSCLC) at Moderate Risk Undergoing Chemotherapy Regimens With Associated Risk Factors
Brief Title: A Study of Efbemalenograstim Alfa Injection for Stage IIIB or IV NSCLC Recieving Moderate-risk Febrile Neutropenia (FN) Chemotherapy Regimen With Risk Factors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUARD-03
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-05

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Lung Cancer; Chemotherapy; Efgbemalenograstim alfa; Absolute Neutrophil Count (ANC) Reduction; Febrile Neutropenia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Febrile Neutropenia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group（primary prevention） (Experimental): Efgbemalenograstim alfa, 20 mg, subcutaneous injection, administered 48±4 hours after the completion of each chemotherapy cycle.
  Interventions: Drug: Efgbemalenograstim alfa
- control group（secondary prevention） (Active Comparator): Efgbemalenograstim alfa, 20 mg, subcutaneous injection, administered 48±4 hours after the completion of the next chemotherapy cycle if ≥ Grade 3 ANC reduction occurs in the preceding chemotherapy cycle.
  Interventions: Drug: Efgbemalenograstim alfa

INTERVENTIONS:
Drug: Efgbemalenograstim alfa — Efbemalenograstim alfa Injection is a recombinant fusion protein composed of the double molecules of human granulocyte colony-stimulating factor (G-CSF) and the Fc fragment of human immunoglobulin (hIgG2). It is used for adult patients with non-myeloid malignancies undergoing myelosuppressive anticancer therapy that is associated with a high risk of febrile neutropenia, to reduce the incidence of infections manifested by febrile neutropenia.

SUMMARY:
The aim of this study was to observe the efficacy and safety of Efbemalenograstim Alfa in the prevention of absolute neutrophil count (ANC) reduction after chemotherapy in NSCLC patients at risk of platinum-containing chemotherapy with risk factors in febrile neutropenia (FN)

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily join this study, sign an informed consent form, exhibit good compliance, and cooperate with follow-up.
2. At the time of signing the informed consent form, participants must be ≥ 18 years old, with no gender restrictions.
3. Stage IIIB-IV NSCLC with negative driver mutations, who have not received chemotherapy or radiotherapy previously.
4. Planned to undergo platinum-based (carboplatin/cisplatin) combined with taxane-based (paclitaxel/albumin-bound paclitaxel/liposomal paclitaxel/paclitaxel polymer micelles) chemotherapy regimen (may be combined with immunotherapy or anti-angiogenic therapy).
5. Have other risk factors related to febrile neutropenia (FN), including but not limited to age ≥65 years, poor nutritional/physical condition (i.e., ECOG score ≥2), etc.
6. Expected survival of at least 12 weeks.
7. Normal function of major organs, meeting the following criteria:

   * Complete blood count criteria (no blood transfusion in the past 14 days, no use of G-CSF or other hematopoietic growth factors for correction):
   * Hemoglobin (Hb) ≥ 90g/L
   * Absolute neutrophil count (ANC) ≥ 2.0×10^9/L
   * Platelets (PLT) ≥ 80×10^9/L
   * Biochemical criteria:
   * Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 ULN
   * Serum creatinine (Cr) ≤ 1.5 ULN or creatinine clearance rate (CrCl) ≥ 50 ml/min
8. Women of childbearing potential must have implemented reliable contraceptive measures or undergone a serum pregnancy test within 7 days before enrollment, with a negative result.
9. Male and female participants of childbearing age must agree to use reliable contraceptive methods from before entering the trial, throughout the study, and for 8 weeks after discontinuation.

Exclusion Criteria:

1. Previously received chemotherapy or radiotherapy, including but not limited to neoadjuvant chemoradiotherapy and/or adjuvant chemoradiotherapy.
2. Underwent bone marrow transplantation or stem cell transplantation.
3. Concurrently diagnosed with malignancies other than NSCLC.
4. Active central nervous system metastasis and/or carcinomatous meningitis, except for asymptomatic brain metastasis subjects (i.e., no progressive central nervous system symptoms caused by brain metastases, no need for corticosteroids, and lesion size ≤1.5 cm) are allowed.
5. Diagnosed with acute congestive heart failure, cardiomyopathy, or myocardial infarction by clinical, electrocardiogram, or other means.
6. Has a disease that may cause splenomegaly.
7. Associated with malignant hematological disorders.
8. Previously experienced sustained Grade ≥3 neutropenia (ANC <1.0×10^9/L) or febrile neutropenia lasting 3 days or more.
9. Underwent surgical procedures within the past 4 weeks and/or has an open wound.
10. Tumor involvement in the bone marrow.
11. Diagnosed with acute infections, chronic active hepatitis B within the past year (unless known negative for hepatitis B virus antigen before selection), or hepatitis C.
12. Pregnant or lactating women.
13. Known positive serum response to human immunodeficiency virus (HIV) or diagnosed with AIDS.
14. Active tuberculosis or recent history of contact with a tuberculosis patient unless tuberculin test is negative; or receiving treatment for tuberculosis; or suspected cases on chest X-ray.
15. Sickle cell anemia.
16. Known allergy to granulocyte colony-stimulating factors or drug excipients.
17. Rubber allergy.
18. Use of other investigational drugs within the past month before enrollment.
19. The investigator believes the participant has a disease or symptoms that make them unsuitable for participation in this study, and the investigational drug may harm the participant's health or affect the judgment of adverse events.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of Grade ≥3 ANC reduction | Up to a year and a half after starting chemotherapy
  The incidence rate of Grade ≥3 ANC reduction during the first chemotherapy cycle for two groups of participants receiving primary and secondary prophylaxis with Efgbemalenograstim alfa in the first treatment cycle.

SECONDARY OUTCOMES:
The incidence rate of FN | Up to a year and a half after starting chemotherapy
  The incidence rate of febrile neutropenia (FN) for each cycle
The incidence rate of Grade ≥3 ANC reduction | Up to a year and a half after starting chemotherapy
  The incidence rate of Grade ≥3 ANC reduction during chemotherapy cycles 2-4/6
Adverse Events | Up to a year and a half after starting chemotherapy
  Including adverse events/serious adverse events and their incidence rates

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - the First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital & Institute, Jinan, Shandong
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: Yes
De-identified individal participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion
Access Criteria: Data access requests will be reviewed by an external indepentent Review Panel. Requesdtors will be required to sign a Data Access Agreement.
URL: http://www.cttq.com/